CLINICAL TRIAL: NCT05574868
Title: Evaluation of the Rigicon Infla10® Three-Piece Inflatable Penile Prosthesis for the Treatment of Patients With Erectile Dysfunction
Brief Title: Rigicon Infla10® Three-Piece Inflatable Penile Prosthesis (ERASE ED)
Acronym: ERASE-ED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGN-ED-IPP-202201
Record Dates: First submitted 2022-10-06; First posted 2022-10-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Erectile Dysfunction
Keywords: Infla10; Rigicon; Dynamic; Erectile Dysfunction; Inflatable Penile Prosthesis; Penile Prosthesis
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Experimental: Rigicon Infla 10® Three-Piece Inflatable Penile Prosthesis Group (Experimental): Male subjects 22 years of age and older who are implanted with an Rigicon Infla 10® Three-Piece Inflatable Penile Prosthesis for erectile dysfunction.
  Interventions: Device: Rigicon Infla 10® Three-Piece Inflatable Penile Prosthesis

INTERVENTIONS:
Device: Rigicon Infla 10® Three-Piece Inflatable Penile Prosthesis — Treatment: Erectile dysfunction
  Other Names: IPP

SUMMARY:
This study evaluates the long-term safety and efficacy of the use of the Rigicon Infla 10® Three-Piece Inflatable Penile Prosthesis in patients with erectile dysfunction. This study follows patients implanted with the Rigicon Infla 10® Three-Piece Inflatable Penile Prosthesis for up to 3 years after implantation.

This study will take approximately 6 months to enroll all subjects. (14 days, 6 weeks, 6 months, 12 months,18 months, 24 months, and 36 months, post-procedure. )

Subjects will be followed per protocol and institutional standard of care for ED and comorbidities.

DETAILED DESCRIPTION:
Erectile dysfunction (ED) is a common male sexual dysfunction associated with a reduced quality of life for patients and their partners. Incidence of ED increases with age and is associated with depression, obesity, diabetes mellitus, hypertension, cardiovascular disease and benign prostatic hyperplasia. ED is diagnosed with symptoms of (1) inability to attain or sustain a penile erection during sexual activity and (2) a reduction of penile rigidity in >75% of sexual encounters during six months period. ED is estimated to affect approximately 52% of men in age of 40 to 70 years.It is projected in 2025, the worldwide ED prevalence of about 322 million. ED usually has organic causes, such as damage of arteries, smooth muscle and fibrous tissue. This resuls in impairment of blood flow to and from penis due to diabetes, renal disease, atherosclerosis and vascular disease.

Management of ED involves in life style modification, medical, surgical interventions, and possibly, in the future, tissue- engineering or cellular or gene therapy. Oral phosphodiesterase type 5 inhibitor (PDE5i), which works with sexual stimulation, is an effective medical therapy for ED with an excellent safety profile. Intracavernosal injection of or topical application vasoactive drug have also been studied. The first inflatable penile prosthesis was introduced in 1973 and current models of inflatable penile prostheses include the AMS 700 series, Coloplast Titan device and Zephyr ZSI device. A patient-activated inflatable penile prosthesis (IPP) provides patients a means to achieve dependable spontaneity for intercourse.

Rigicon has developed a three-piece inflatable penile prosthesis (IPP) (Infla10®) for the treatment of ED. This proposed study is to assess the safety and effectiveness of the Rigicon IPP in treating ED. Clinical literature and preclinical testing, including biocompatibility, device validation and verification, and animal studies support the safety and efficacy of this device for the intended therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥22 years of age.
2. Diagnosed with erectile dysfunction (impotence).
3. Agree to receive Infla10® three-piece IPP as an ED treatment.
4. Willing to complete all protocol required follow-up visits and tests.

Exclusion Criteria:

1. 1. Contraindication to general anesthesia.
2. Known allergy or sensitivity to product materials as indicated in the device labeling.
3. Previous penile prosthesis or prior enlargement surgeries
4. Diagnosed penile sensory neuropathy.
5. Diagnosed with fibrotic disease, such as priapism, Peyronie's disease or Chordee.
6. Compromised immune system, such as systemic lupus erythematosus, discoid lupus, or scleroderma
7. Patients who are receiving immunosuppressive drugs or have a history of kidney transplantation
8. Uncontrolled diabetes (Fasting Blood Sugar FBS) >300 or HbA1c ≥9.0 on morning of surgery)
9. Bleeding disorder or coagulopathy that may in the judgment of the investigator preclude safe procedure.
10. Active urogenital infection or active skin infection in region of surgery or systemic infection at the time of assessment.
11. Clinically significant comorbidities or presence of unstable conditions (e.g. cardiovascular, lung, renal [serum creatinine > 2.0 mg/dl], hepatic, bleeding disorders, or metabolic impairment) that may confound the results of the study or in the judgment of the physician investigator preclude safe procedure.
12. Any cognitive disorder that interferes with or precludes direct and accurate communication with the study investigator regarding the study or affects the ability to complete the study questionnaires.
13. Lacking manual dexterity or mental abilities necessary to operate the device.
14. Expected life expectancy < two years.
15. Unwilling or unable to sign the Informed Consent.
16. Unwilling or unable to comply with the follow-up study requirements.
17. Currently participating in an investigational drug or another investigational device exemption (IDE) study.
18. Incarcerated subjects
19. Psychogenic erectile dysfunction

Min Age: 22 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 182 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2026-05-21 (Estimated); Study Completion 2026-05-21 (Estimated)

PRIMARY OUTCOMES:
The primary safety outcome is the proportion of participants free from any device- or procedure-related adverse event of CTCAE Grade ≥2 through 12 months post-procedure, graded per CTCAE v5.0 and IPP-specific mapping. | 12 months
  Description: Success will be concluded if the two-sided 95 percent confidence interval (equivalently, one-sided 97.5 percent) for the 12-month proportion has its lower bound strictly greater than 0.90 as specified in the statistical plan.
The primary effectiveness endpoint is a binary "pass" or "fail" objective axial rigidity test, assessed at 12 months. | 12 months
  Description: The objective axial rigidity test will use a calibrated axial-rigidity device to measure vertical displacement of the fully inflated penis under a standardized 650-gram load. ≤15 mm displacement will be counted as a "pass". Success will be concluded if the two-sided 95 percent confidence interval for the 12-month success proportion has its lower bound strictly greater than the pre-specified performance goal in the statistical plan.

SECONDARY OUTCOMES:
Durability | 12 months
  Description: A secondary durability endpoint will summarize "revision- or explant-free survival" using Kaplan-Meier methods, with participants without an event right-censored at last contact.
International Index of Erectile Function - Erectile Function (IIEF-EF) Domain Score | Baseline (pre-implantation) and Months 3, 6, 12, 18, 24, and 36 post-implantation.
  The Erectile Function (EF) domain of the IIEF-15 questionnaire (Items 1-5 and 15) will be used to assess patient erectile function. Change from baseline in the EF domain total score will be reported at each time point. The questionnaire may be completed remotely via ePRO.
  Scale / Range: 6-30 points Direction: Higher scores indicate better erectile function. Assessment Schedule: Baseline and Months 3, 6, 12, 18, 24, and 36.
Rosenberg Self-Esteem Scale (RSES) Total Score | Baseline (pre-implantation) and Months 3, 6, 12, 18, 24, and 36 post-implantation.
  The 10-item Rosenberg Self-Esteem Scale (RSES) is a validated self-report instrument used to measure global self-worth by assessing positive and negative feelings about the self. The total RSES score will be used as a secondary endpoint to evaluate change in participant self-esteem and psychosocial well-being following device implantation.
  Administration and scoring: Each item is rated on a 4-point Likert scale (1 = Strongly Disagree to 4 = Strongly Agree). Items 2, 5, 6, 8, and 9 are reverse scored. The total score ranges from 10 to 40, with higher scores indicating greater self-esteem.
  Analysis: Change from baseline in total RSES score will be summarized at each time point as mean ± standard deviation with 95% confidence intervals, and formally tested within the pre-specified hierarchical secondary endpoint sequence.
  Scale / Range: 10-40 points Direction: Higher scores indicate higher self-esteem (better outcome).

OTHER OUTCOMES:
Adverse Events | 36 months
  Description: Descriptive tabulations by system organ class and preferred term, including device-relatedness and seriousness, and rates for typical post-IPP events categorized as AEs, SAEs, and UADEs.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Love, Dr., Principal Investigator — Urology South at Holmesglen Private Hospital; Boon K. Kua, Dr., Study Director — Wesley Hospital; Hodo Haxhimolla, Dr., Study Director — Canberra Laparoscopic, Robotic & Laser Urology Centre; Phillip Katelaris, Dr., Study Director — Katelaris Urology; William Lynch, Dr., Study Director — St George Urology; Steven Wilson, Dr., Study Director — Department of Urology, Institute for Urologic Excellence; Paul Perito, MD, Study Director — Perito Urology - Penile Implant Clinic; Gerard Testa, Dr., Study Director — Shire Urology; Daniel Moon, Dr., Study Director — Advanced Urology Melbourne
Locations (7):
- Australia (7):
  - Wesley Hospital, Auchenflower
  - Canberra Laparoscopic, Robotic & Laser Urology Centre, Garran
  - Katelaris Urology, Hornsby
  - St George Urology, Hurstville
  - Advanced Urology Melbourne, Malvern
  - Shire Urology, Miranda
  - Urology South at Holmesglen Private Hospital, Moorabbin

IPD SHARING:
Plan to Share IPD: No